CLINICAL TRIAL: NCT06121154
Title: A Possible Association Between Pseudoexfoliation Syndrome, Sarcopenia and Chronic Pain
Brief Title: Pseudoexfoliation Syndrome, Sarcopenia and Chronic Pain
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Onur Armağan, Prof., Eskisehir Osmangazi University
Other Study IDs: SarcoPEX
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Sarcopenia; Pseudoexfoliation Syndrome
Keywords: sarcopenia; pseudoexfoliation syndrome; chronic pain
MeSH Terms: conditions — Sarcopenia; Exfoliation Syndrome; Chronic Pain | interventions — Walking Speed; Hand Strength; Visual Analog Scale

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEX-positive patients: The criteria to diagnose Pseudoexfoliation syndrome (PEX) were, after pupillary dilatation, the presence of white fluffy dandruff-like material on one or more anterior segment structures, including the pupillary margin, the anterior lens capsule, or the angle in biomicroscopic examination. The patients were divided into two groups: solely based on PEX-positive (n=48) and PEX-negative (n=48) status
  Interventions: Diagnostic Test: SARC-F questionnaire; Diagnostic Test: Gait speed; Diagnostic Test: The chair rise test; Diagnostic Test: Grip strength; Diagnostic Test: Visual analog scale
- PEX-negative patients: The criteria to diagnose Pseudoexfoliation syndrome (PEX) were, after pupillary dilatation, the presence of white fluffy dandruff-like material on one or more anterior segment structures, including the pupillary margin, the anterior lens capsule, or the angle in biomicroscopic examination. The patients were divided into two groups: solely based on PEX-positive (n=48) and PEX-negative (n=48) status
  Interventions: Diagnostic Test: SARC-F questionnaire; Diagnostic Test: Gait speed; Diagnostic Test: The chair rise test; Diagnostic Test: Grip strength; Diagnostic Test: Visual analog scale

INTERVENTIONS:
Diagnostic Test: SARC-F questionnaire — The SARC-F scale has 5 questions which evaluate strength, assistance in ambulation, rising from a chair, stair climbing, and falls. The cut off point for predicting sarcopenia is score 4; "4 and more" means risk of sarcopenia.
Diagnostic Test: Gait speed — Low gait speed was defined as walking below than 0.8 meters per second.
Diagnostic Test: The chair rise test — the chair rise test (measures the strength of leg muscles), it measures the time taken for 5 times of rising from the sitting position without using arms, and was defined as low when the time taken was more than 15 seconds
Diagnostic Test: Grip strength — Grip strength was measured with a hand-held dynamometer (Baseline, White Plains, New York, USA), and the cut-off thresholds were 32 kg for males and 22 kg for females
Diagnostic Test: Visual analog scale — The visual analogue scale (VAS) was used for measuring general body pain severity, which was assessed from 0 (no pain) to 10 (worst possible pain)

SUMMARY:
Aim: Pseudoexfoliation syndrome (PEX) is a systemic disease of connective tissue, it can also contribute to sarcopenia and chronic musculoskeletal pain with common pathways.

1. First aim of this study was to investigate whether the rate of sarcopenia is higher in patients with PEX
2. Second aim was to investigate the association between PEX, sarcopenia parameters and chronic musculoskeletal pain.

Methods: A total of 96-patients were enrolled in this study and divided into two groups: PEX-positive (n=48) and PEX-negative (n=48) patients. The variables: the demographic data, sarcopenia parameters (SARC-F-questionnaire, hand-grip strength, chair-rise test, gait speed) and pain parameters (having any chronic musculoskeletal pain, pain regions and visual analogue scale-pain).

DETAILED DESCRIPTION:
Sarcopenia is defined as a decreased muscle mass, muscle strength and muscle function, which leads to lower physical performance, disability and quality of life. Pseudoexfoliation syndrome (PEX) is an age-related, genetic and systemic disease characterized by the accumulation of abnormal extracellular fibrillar material in many ocular and extraocular tissues Aim: Pseudoexfoliation syndrome (PEX) is a systemic disease of connective tissue, it can also contribute to sarcopenia and chronic musculoskeletal pain with common pathways.

1. First aim of this study was to investigate whether the rate of sarcopenia is higher in patients with PEX
2. Second aim was to investigate the association between PEX, sarcopenia parameters and chronic musculoskeletal pain.

Methods: A total of 96-patients were enrolled in this study and divided into two groups according to having pseudoexfoliation material in ocular tissues: PEX-positive (n=48) and PEX-negative (n=48) patients. The variables: the demographic data, sarcopenia parameters (SARC-F-questionnaire, hand-grip strength, chair-rise test, gait speed) and pain parameters (having any chronic musculoskeletal pain, pain regions and visual analogue scale-pain).

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years

  * Undergoing a detailed complete ophtalmic examination by an experienced physician within 1 month at the Department of Ophtalmology in the same university hospital.

Exclusion Criteria:

* having ophtalmic diseases that cause vision loss and reduce quality of life and mobility smoking, acute/subacute pain, amputation, infection, active arthritis, active cancer, having any protesis or surgery in lower extremities and low back, neurological disorders, malabsorption, weight loss, uncontrolled major systemic diseases, impaired cognitive function and being immobilised.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case-control study was conducted with 98 patients who admitted to Department of Physical Medicine and Rehabilitation Outpatient Clinic, Eskişehir Osmangazi University Hospital between March-August 2023.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
SARC-F | Baseline
  The SARC-F scale has 5 questions which evaluate strength, assistance in ambulation, rising from a chair, stair climbing, and falls. The cut off point for predicting sarcopenia is score 4; "4 and more" means risk of sarcopenia.

SECONDARY OUTCOMES:
Grip strength | Baseline
  Grip strength was measured with a hand-held dynamometer (Baseline, White Plains, New York, USA), and the cut-off thresholds were 32 kg for males and 22 kg for females
Visual analog scale | Baseline
  The visual analogue scale (VAS) was used for measuring general body pain severity, which was assessed from 0 (no pain) to 10 (worst possible pain)
The chair rise test | Baseline
  It measures the time taken for 5 times of rising from the sitting position without using arms, and was defined as low when the time taken was more than 15 seconds
Gait speed | Baseline
  Low gait speed was defined as walking below than 0.8 meters per second.

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Assoc Prof, Study Director — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No